CLINICAL TRIAL: NCT01227265
Title: A Phase 3, 12 Week, Double-blind, Placebo-controlled Efficacy and Safety Study of Preladenant in Subjects With Moderate to Severe Parkinson's Disease.
Brief Title: Placebo Controlled Study of Preladenant in Participants With Moderate to Severe Parkinson's Disease (P07037)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P07037; 2010-020112-11 (EudraCT Number); MK-3814-028 (Other: Merck Study Number)
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Results first posted 2016-04-12 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-08

CONDITIONS: Parkinson Disease; Idiopathic Parkinson Disease; Idiopathic Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — 2-(2-furanyl)-7-(2-(4-(4-(2-methoxyethoxy)phenyl)-1-piperazinyl)ethyl)-7H-pyrazolo(4,3-e)(1,2,4)triazolo(1,5-c)pyrimidine-5-amine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Preladenant 2 mg (Experimental): Participants received 2 mg as a single oral dose twice daily for 12 weeks. Participants could then enroll in an extension trial or return for a follow-up visit two (2) weeks later.
  Interventions: Drug: Preladenant
- Preladenant 5 mg (Experimental): Participants received 5 mg as a single oral dose twice daily for 12 weeks. Participants could then enroll in an extension trial or return for a follow-up visit two (2) weeks later.
  Interventions: Drug: Preladenant
- Placebo (Placebo Comparator): Participants received preladenant-matching placebo as a single oral dose twice daily for 12 weeks. Participants could then enroll in an extention trial or return for a follow-up visit two (2) weeks later.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Preladenant — Preladenant 2 mg or 5 mg oral tablet taken twice daily
  Other Names: SCH 420814; MK-3814
  Arms: Preladenant 2 mg; Preladenant 5 mg
Drug: Placebo — Preladenant-matching placebo oral tablet taken twice daily
  Arms: Placebo

SUMMARY:
This is a study of the efficacy and safety of preladenant in adult participants with moderate to severe Parkinson's Disease (PD). While on this study, participants will continue to take their usual, prescribed, stable regimen of levodopa (L-dopa) or L-dopa plus adjunct PD medications and will be randomized to receive 2 mg preladenant, 5 mg preladenant, or placebo, twice daily, for 12 weeks. After that, participants may choose to receive additional treatment with preladenant. The primary hypothesis is that at least the 5 mg twice daily dose of preladenant is superior to placebo as measured by the change from Baseline to Week 12 in the mean "off" time.

ELIGIBILITY:
Inclusion Criteria:

* Each participant must have a diagnosis of idiopathic Parkinson's disease.
* Each participant must have received prior therapy with L-dopa for approximately 1 or more years immediately before Screening and must continue to have a beneficial clinical response to L-dopa.
* Each participant must have been on a stable dopaminergic treatment regimen for at least the 5 weeks immediately before Randomization. Participants receiving other adjunctive treatments (eg, dopamine agonist, anticholinergics) are permitted to enroll in this trial. Participants taking only L-dopa are permitted to enroll in this trial.
* Each participant must be experiencing motor fluctuations with or without dyskinesias within the 4 weeks immediately before Screening, must be experiencing a minimum of 2 hours/day of "off" time, and have a Hoehn & Yahr stage between 2.5 and 4 when in the "on" state.
* Each participant, with or without the help of a caregiver, must be capable of maintaining an accurate and complete symptom diary and to adhere to dose and visit schedules.
* Each participant must have results of Screening clinical laboratory tests drawn within 5 weeks prior to Randomization clinically acceptable to the investigator and not within the parameters specified for exclusion (below).
* All participants who are sexually active or plan to be sexually active agree to use a highly effective method of birth control while in the study and for 2 weeks after the last dose of study drug. A male participant must also not donate sperm within 2 weeks after the last dose of study drug.

Exclusion Criteria:

* A participant must not have a form of drug induced or atypical parkinsonism, a cognitive impairment, bipolar disorder, untreated major depressive disorder, schizophrenia, or other psychotic disorder; history exposure to a known neurotoxin, or any neurological features not consistent with the diagnosis of PD as assessed by the investigator.
* A participant must not have a history of repeated strokes or head injuries, or a stroke within 6 months of Screening; poorly controlled diabetes; abnormal renal function; or a severe or ongoing unstable medical condition.
* A participant must not have had surgery for their PD.
* A participant must not be at imminent risk of self-harm or harm to others.
* A participant must not have a systolic blood pressure (BP) ≥150 mm Hg OR diastolic BP ≥95 mm Hg at Screening and at 2 BP rechecks prior to study start.
* A participant must not have had any clinically significant cardiovascular event or procedure for 6 months prior to study start, including, but not limited to, myocardial infarction, angioplasty, unstable angina, or heart failure; and a participant must not have heart failure staged New York Heart Association Class III or IV.
* A participant must not have an alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥3 x the upper limit of normal (ULN) or total bilirubin (T BIL) ≥1.5 x ULN.
* A participant must not have a history of serologically confirmed hepatic dysfunction (defined as viral infection [Hepatitis B, C, or E; Epstein-Barr virus (EBV); cytomegalovirus (CMV)]) or a history of diagnosis of drug- or alcohol- induced hepatic toxicity or frank hepatitis.
* A participant must not have a history within the past 5 years of a primary or recurrent malignant disease with the exception of adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or in situ prostate cancer with a normal prostate-specific antigen (PSA) post resection.
* A participant must not have received certain prespecified medications for a prespecified time window before the trial.
* A participant must not have an average daily consumption of more than three 4 ounce glasses (118 mL) of wine or the equivalent.
* A participant must not have a severe or ongoing unstable medical condition (eg, any form of clinically significant cardiac disease, symptomatic orthostatic hypotension, seizures, or alcohol/drug dependence).
* A participant must not have allergy/sensitivity to investigational product(s) or its/their excipients.
* A participant must not be breast-feeding, considering breast-feeding, pregnant, or intending to become pregnant.
* A participant must not have used preladenant ever, or any investigational drugs within 90 days immediately before Screening.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2010-11-19 (Actual); Primary Completion 2013-04-04 (Actual); Study Completion 2013-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Hauser RA, Stocchi F, Rascol O, Huyck SB, Capece R, Ho TW, Sklar P, Lines C, Michelson D, Hewitt D. Preladenant as an Adjunctive Therapy With Levodopa in Parkinson Disease: Two Randomized Clinical Trials and Lessons Learned. JAMA Neurol. 2015 Dec;72(12):1491-500. doi: 10.1001/jamaneurol.2015.2268. PMID 26523919

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants with a diagnosis of moderate to severe idiopathic Parkinson's disease were selected to participate in this study.
Pre-assignment Details: After a Screening Period of up to 5 weeks, participants were randomized into 1 of 3 treatment groups (preladenant 2 or 5 mg twice daily or placebo) for 12 weeks. At the end of treatment, participants could choose to enter into an extension trial or return for a follow-up visit 2 weeks later.
Period: Overall Study
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Placebo
Started | 158 | 159 | 159
Treated | 157 | 157 | 159
Completed | 139 | 139 | 145
Not Completed | 19 | 20 | 14
Not completed — Did Not Receive Treatment | 1 | 2 | 0
Not completed — Administrative | 1 | 0 | 2
Not completed — Did Not Meet Protocol Eligibility | 0 | 0 | 1
Not completed — Protocol Violation | 2 | 1 | 0
Not completed — Withdrawal by Subject | 7 | 7 | 3
Not completed — Lost to Follow-up | 2 | 0 | 3
Not completed — Adverse Event | 6 | 10 | 5

BASELINE CHARACTERISTICS:
Population: All Participants as Treated - all participants who received at least one dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Placebo | Total
Number analyzed (Participants) | 157 | 157 | 159 | 473
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.9 (9.0) | 64.2 (8.7) | 64.2 (8.9) | 63.8 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 71 | 64 | 184
  Male | 108 | 86 | 95 | 289

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average "Off" Time (Hours Per Day) at Week 12
Description: The "on" state is defined as the period of time during which a patient's symptoms of PD improve or disappear following treatment with L-dopa or dopamine agonists. The "off" state is defined as the period of time characterized by the return of symptoms (i..e. tremor, slowness, and rigidity) following treatment with L-dopa or dopamine agonists. Study participants reported their symptoms at half-hour intervals as "off", "on", or "asleep" on their daily diary for 3 days before randomization (baseline) and for the 3 days immediately before their Week 12 visit. The mean change from baseline in "off" time was based on a constrained longitudinal data analysis (cLDA) with treatment, time, and treatment-by-time interaction as fixed effects and subject as random effect.
Time Frame: Baseline and Week 12
Population: Full Analysis Set (FAS): All randomized participants remaining after participants were excluded for failure to receive at least one dose of study treatment, lack of any post-randomization endpoint data subsequent to at least 1 dose of study treatment, or lack of Baseline data for those analyses requiring Baseline data.
Measure: Mean (Standard Error); unit: hours per day
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Placebo
Number analyzed (Participants) | 154 | 153 | 158
hours per day | -1.0 (0.20) | -1.1 (0.20) | -0.8 (0.19)
Statistical Analysis 1: Comparison: Preladenant 2 mg vs Placebo; Test type: Superiority or Other; p = 0.4933, cLDA; Difference in Estimated Means = -0.2, 95% CI 2-sided [-0.72 to 0.35]
Statistical Analysis 2: Comparison: Preladenant 5 mg vs Placebo; Test type: Superiority or Other; p = 0.2364, cLDA; Difference in Estimated Means = -0.3, 95% CI 2-sided [-0.86 to 0.21]

2. Secondary Outcome: Percentage of Participants With >30% Change (Reduction) From Baseline at Week 12 in Mean "Off" Time
Description: A participant with at least a 30% reduction in mean "off" time from Baseline to End of Treatment (Week 12) is considered as "responder". The "on" state is defined as the period of time during which a patient's symptoms of PD improve or disappear following treatment with L-dopa or dopamine agonists. The "off" state is defined as the period of time characterized by the return of symptoms (i..e. tremor, slowness, and rigidity) following treatment with L-dopa or dopamine agonists. Study participants reported their symptoms at half-hour intervals as "off", "on", or "asleep" on their daily diary for 3 days before randomization and for the 3 days immediately before their Week 12 visit.
Time Frame: Baseline and Week 12
Population: Full Analysis Set (FAS): All randomized participants remaining after participants were excluded for failure to receive at least one dose of study treatment, lack of any post-randomization endpoint data subsequent to at least one dose of study treatment, or lack of Baseline data for those analyses requiring Baseline data.
Measure: Number; unit: Percentage of participants
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Placebo
Number analyzed (Participants) | 154 | 153 | 158
Percentage of participants | 37.1 | 36.9 | 30.5
Statistical Analysis 1: Comparison: Preladenant 2 mg vs Placebo; Test type: Superiority or Other; p = 0.244, Mixed Models Analysis — p-value is for the estimated Odds Ratio based on a generalized linear mixed model with baseline average OFF time (hours/day) as a covariate and treatment-by-time interaction as fixed effect and participant as random effect; Estimated Difference in Percentage = 7.0, 95% CI 2-sided [-4.17 to 18.05]
Statistical Analysis 2: Comparison: Preladenant 5 mg vs Placebo; Test type: Superiority or Other; p = 0.262, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Estimated Difference in Percentage = 6.5, 95% CI 2-sided [-4.63 to 17.61]

3. Secondary Outcome: Change From Baseline in Average "On" Time (Hours Per Day) Without Troublesome Dyskinesia at Week 12
Description: "On" time is when a PD participant's symptoms are improved. Mean "on" time without troublesome dyskinesias is derived from the available diary data collected for 3 days immediately prior to a clinic visit. "On" time without troublesome dyskinesia is the sum of "on" time without dyskinesia plus "on" time with non-troublesome dyskinesia as recorded in the diary. The mean change from baseline in "on" time was based on a cLDA with treatment, time, and treatment-by-time interaction as fixed effects and subject as random effect.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: hours per day
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Placebo
Number analyzed (Participants) | 154 | 153 | 158
hours per day | 0.6 (0.21) | 0.7 (0.21) | 0.5 (0.20)
Statistical Analysis 1: Comparison: Preladenant 2 mg vs Placebo; Test type: Superiority or Other; p = 0.776, cLDA; Difference in Estimated Means = 0.1, 95% CI 2-sided [-0.47 to 0.63]
Statistical Analysis 2: Comparison: Preladenant 5 mg vs Placebo; Test type: Superiority or Other; p = 0.683, cLDA; Difference in Estimated Means = 0.1, 95% CI 2-sided [-0.44 to 0.67]

4. Primary Outcome: Number of Participants With Systolic Blood Pressure (SBP) ≥180 mmHg and 20 mmHg Increase
Description: The number of participants with Systolic Blood Pressure (SBP) ≥180 mmHg and 20 mmHg increase was reported. Participants lie supine at rest for 5 minutes, then have a single BP measurement taken (ie, 1 reading). Participants then stand for 3 minutes at rest, followed by a single BP measurement (1 reading) in the standing position.
Time Frame: Up to Week 14
Population: All Participants as Treated (APaT): All participants who received at least one (1) dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Placebo
Number analyzed (Participants) | 157 | 157 | 159
Participants
  Supine | 0 | 1 | 0
  Standing | 1 | 0 | 0

5. Primary Outcome: Number of Participants With Diastolic Blood Pressure (DBP) ≥105 mmHg and 15 mmHg Increase
Description: The number of participants with Diastolic Blood Pressure (DBP) ≥105 mmHg and 15 mmHg increase was reported. Participants lie supine at rest for 5 minutes, then have a single BP measurement taken (ie, 1 reading). Participants then stand for 3 minutes at rest, followed by a single BP measurement (1 reading) in the standing position.
Time Frame: Up to Week 14
Population: All Participants as Treated (APaT): All participants who received at least one (1) dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Placebo
Number analyzed (Participants) | 157 | 157 | 159
Participants
  Supine | 1 | 2 | 3
  Standing | 7 | 3 | 6

6. Primary Outcome: Percentage of Participants With Suicidality
Description: The percentage of participants with suicidality using the Columbia - Suicide Severity Rating Scale (C-SSRS) was reported. The C-SSR was used in this study only for the purpose of safety monitoring by measuring the incidence of different types of suicidality categories during treatment. The assessment was done by the nature of the responses, not by a numbered scale. Participants who reported at least one occurrence of suicidal behavior or suicidal ideation were counted as having experienced suicidality. Suicidal behavior included suicide attempt, aborted attempt, interrupted attempt, or preparatory behavior. Suicidal ideation included a wish to die or active suicidal thought with or without method, intent or plan.
Time Frame: Up to Week 12
Population: All Participants as Treated (APaT): All participants who received at least one (1) dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Placebo
Number analyzed (Participants) | 157 | 157 | 159
Percentage of participants | 3 | 4 | 1

7. Primary Outcome: Change From Baseline in Total Epworth Sleepiness Scale (ESS) at Week 12
Description: The ESS is a self-administered questionnaire providing a measure of a person's general level of daytime sleepiness, or their average sleep propensity in daily life. The scale consists of 8 situations in which the participant rates their tendency to become sleepy on a scale of 0=no chance of dozing to 3=high chance of dozing. The overall score is the sum of the scores for the 8 situations for a minimum of 0 and a maximum of 24 with a higher score indicating greater sleepiness. The mean change from baseline in total EES was based on a cLDA with treatment, time, and treatment-by-time interaction as fixed effects and subject as random effect.
Time Frame: Baseline and Week 12
Population: All Participants as Treated (APaT): All participants who received at least one (1) dose of study drug.
Measure: Mean (Standard Error); unit: Score on a Scale
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Placebo
Number analyzed (Participants) | 157 | 157 | 159
Score on a Scale | -0.4 (0.28) | -0.0 (0.29) | -0.2 (0.28)
Statistical Analysis 1: Comparison: Preladenant 2 mg vs Placebo; Test type: Superiority or Other; p = 0.6968, cLDA; Difference in Estimated Means = -0.2, 95% CI 2-sided [-0.92 to 0.61]
Statistical Analysis 2: Comparison: Preladenant 5 mg vs Placebo; Test type: Superiority or Other; p = 0.6142, cLDA; Difference in Estimated Means = 0.2, 95% CI 2-sided [-0.57 to 0.97]

ADVERSE EVENTS:
Time Frame: Up to 14 weeks (including 14 days of follow-up)
Description: All Participants as Treated
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 5/157 | 2/157 | 4/159
Other Adverse Events (participants affected / at risk) | 37/157 | 46/157 | 25/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preladenant 2 mg (N=157) | Preladenant 5 mg (N=157) | Placebo (N=159)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Kidney Rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wrist Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral Haematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Completed Suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Stress Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preladenant 2 mg (N=157) | Preladenant 5 mg (N=157) | Placebo (N=159)
Constipation (Gastrointestinal disorders) | 11 (11) | 15 (18) | 4 (4)
Nausea (Gastrointestinal disorders) | 5 (6) | 9 (10) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 7 (9) | 9 (12) | 10 (14)
Dizziness (Nervous system disorders) | 10 (11) | 6 (6) | 3 (3)
Dyskinesia (Nervous system disorders) | 3 (3) | 11 (13) | 5 (5)
Headache (Nervous system disorders) | 12 (13) | 10 (11) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial.